CLINICAL TRIAL: NCT04230265
Title: Multicenter, Open-label, Adaptive Design Phase I Trial With Genetically Modified T-cells Carrying Universal Chimeric Antigen Receptors (UniCAR02-T) in Combination With CD123 Target Module (TM123) for the Treatment of Patients With Hematologic and Lymphatic Malignancies Positive for CD123
Brief Title: Phase 1 Study of UniCAR02-T-CD123 in Patients With Selected CD123 Positive Hematologic Malignancies
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: business decision by sponsor
Sponsor: AvenCell Europe GmbH (Industry)
Collaborators: PHARMALOG Institut für klinische Forschung GmbH (Unknown)
Responsible Party: Sponsor
Organization: AvenCell Therapeutics, Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UC02-123-01; 2019-001339-30 (EudraCT Number); 2024-515827-12-00 (EU CTIS Number)
Record Dates: First submitted 2020-01-10; First posted 2020-01-18 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Acute Myeloid Leukemia (AML)
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — Cyclophosphamide; fludarabine; Inosine Monophosphate

STUDY DESIGN:
Intervention Model Description: Phase 1b Dose Expansion: An expansion cohort of up to 20 patients was initiated.
Masking Description: In the expansion cohort 2 different TM123 dose levels shall be compared descriptively.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- UniCAR02-T-CD123 (4 mg/day TM123) (Experimental): Preconditioning (lymphodepletion) with cyclophosphamide and fludarabine, followed by combination treatment of genetically modified T-cells carrying universal chimeric antigen receptors (UniCAR02-T) with 4 mg/day of the recombinant antibody derivative TM123.
  Interventions: Drug: Cyclophosphamide (Non-IMP); Drug: Fludarabine (Non-IMP); Drug: TM123 (IMP); Drug: UniCAR02-T (IMP)
- UniCAR02-T-CD123 (8 mg/day TM123) (Experimental): Preconditioning (lymphodepletion) with cyclophosphamide and fludarabine, followed by combination treatment of genetically modified T-cells carrying universal chimeric antigen receptors (UniCAR02-T) with 8 mg/day of the recombinant antibody derivative TM123.
  Interventions: Drug: Cyclophosphamide (Non-IMP); Drug: Fludarabine (Non-IMP); Drug: TM123 (IMP); Drug: UniCAR02-T (IMP)

INTERVENTIONS:
Drug: Cyclophosphamide (Non-IMP) — Intravenous infusion over 3 days
Drug: Fludarabine (Non-IMP) — Intravenous infusion over 3 days
Drug: TM123 (IMP) — Intravenous Infusion for 20 days
Drug: UniCAR02-T (IMP) — Intravenous infusion of single dose

SUMMARY:
This dose-escalating phase I trial assesses for the first time the safety, the side effects and the harmlessness, as well as the therapeutical benefit of the new study drug UniCAR02-T-CD123 in patients with hematologic and lymphatic malignancies positive for CD123 marker. The UniCAR02-T-CD123 drug is a combination of a cellular component (UniCAR02-T) with a recombinant antibody derivative (TM123) which together forms the active drug.

ELIGIBILITY:
Phase 1a Dose Escalation:

Inclusion Criteria:

1. Male or female patients, age ≥ 18 years
2. Documented definitive diagnosis of Relapsed or refractory AML (according to standard of care testing) and CD123 positivity of ≥20 % of blasts. MRD+ AML without morphological relapse or refractoriness may be included with the sponsor's approval
3. Eastern Cooperative Oncology Group (ECOG) of 0 to 1
4. Life expectancy of at least 2 months
5. Adequate renal and hepatic laboratory assessments
6. Adequate cardiac function
7. Long-term venous access existing (e.g. port-system) resp. acceptance of implantation of a device
8. Able to give written informed consent
9. Weight ≥ 45 kg
10. Negative pregnancy test; routinely using a highly effective method of birth control

Exclusion Criteria:

1. Acute promyelocytic leukemia
2. AML with only extramedullary manifestations (e.g., chloroma, primary myeloid sarcoma).
3. Refractory disease under anti-leukemic treatment lasting longer than 6 months
4. Current manifestation of AML in central nervous system
5. Bone marrow failure syndromes (e.g. Fanconi anemia, Kostman syndrome, Shwachman syndrome)
6. Significant cardiac disease: i.e., heart failure (NYHA III or IV); unstable coronary artery disease, myocardial infarction or serious cardiac ventricular arrhythmias requiring anti-arrhythmic therapy within the last 12 months prior to study entry that may in the Investigator's opinion interfere with participation in the trial.
7. Patients undergoing renal dialysis
8. Pulmonary disease with clinically relevant hypoxia
9. Parkinson's disease, epilepsy, stroke, seizures, significant paresis or aphasia with clinical symptoms in the previous 12 months that may in the Investigator's opinion interfere with participation in the trial.
10. Disseminated intravascular coagulation (DIC) within 3 months prior to the planned start of the study treatment.
11. Hemorrhagic cystitis
12. Active infectious disease considered by investigator to be incompatible with protocol or being contraindications for lymphodepletion therapy
13. Allogeneic stem cell transplantation within last two months or GvHD requiring systemic immunosuppressive therapy
14. Vaccination with live viruses within 2 weeks prior to lymphodepletion therapy
15. Major surgery within 28 days (prior to start of TM123 infusion)
16. Other malignancy requiring active therapy, but adjuvant endocrine therapy is allowed
17. Treatment with any investigational drug substance or experimental therapy within 4 weeks or 5 half-lives (whatever is shorter) of the substance prior to the day of apheresis
18. Prior treatment with gene therapy products unless approved by the sponsor
19. Use of checkpoint inhibitors within 5 half-lives of the respective substance
20. Pregnant or breastfeeding women
21. Currently significant psychologic disorder, including substance abuse
22. Known history of human immunodeficiency virus (HIV) or human T-lymphotropic virus (HTLV) or active/chronic infection with hepatitis C virus (HCV) or hepatitis B virus (HBV)
23. Any significant autoimmune disease requiring systemic immunosuppressive therapy or that may otherwise, in the Investigator's opinion, interfere with participation in the trial, or documented presence of autoantibodies against La/SS-B.

Phase 1b Dose Expansion:

Inclusion Criteria:

1. Male or female patients, age ≥ 18 years
2. Relapsed or refractory AML (according to standard of care testing), having up to 30% blasts in a bone marrow assessment at either screening or prescreening, or patients having between 30% and 40% blasts for 2 consecutive bone marrow assessments with a minimum of 1 months and no more than 2 months apart, and without hyperproliferative disease requiring cytoreductive treatment, up to 3rd relapse, without further approved curative or life-extending treatment options, and documented CD123 positivity of ≥ 20 % of blasts. Exceptions to BM blast criterion are only possible in minor deviations in timing and/or blast count in clinically stable patients, and only with written sponsor approval. Exemptions to CD123 expression are not allowed. MRD+ AML without morphological relapse or refractoriness may be included with the sponsor's approval.
3. Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 1
4. Life expectancy of at least 2 months
5. Adequate renal and hepatic laboratory assessments:

   1. Aspartate aminotransferase (AST), alanine aminotransferase (ALT) and alkaline phosphatase (ALP) ≤ 2.5× upper limit of normal (ULN)
   2. Total bilirubin ≤ 1.5× ULN
   3. Serum creatinine clearance at least 70 mL/min)
6. Adequate cardiac function, i.e., left ventricular ejection fraction (LVEF) of ≥ 50 %.
7. Long-term venous acces existing (e.g., port-system) resp. acceptance of implantation of a device
8. Able to give written informed consent
9. Weight ≥ 45kg
10. Negative pregnancy test; routinely using a highly effective method of birth control

    Exclusion criteria:
11. Acute promyelocytic leukemia (t15;17)
12. AML with only extramedullary manifestations (e.g., chloroma, primary myeloid sarcoma)
13. Refractory disease under anti-leukemic treatment lasting longer than 6 months
14. Current manifestion of AML in central nervous system
15. Bone marrow failure syndromes (e.g. Fanconi anemia, Kostman syndrome, Schwachman syndrome)
16. Significant cardiac disease: i.e., heart failure (NYHA III or IV); unstable coronary artery disease, myocardial infarction or serious cardiac ventricular arrhythmias requiring anti-arrhythmic therapy within the last 12 months prior to study entry that may in the Investigator''s opinion interfere with participation in the trial.
17. Patients undergoing renal dialysis
18. Pulmonary disease with clinically relevant hypoxia
19. Parkinson's disease, epilepsy, stroke, seizures, significant paresis or aphasia with clinical symptoms in the previous 12 months that may in the Investigator's opinion interfere with participation in the trial.
20. Disseminated intravascular coagulation (DIC) within 3 months prior to the planned start of the study treatment.
21. Hemorrhagic cystitis
22. Active infections disease considered by investigator to be incompatible with protocol or being contraindications for lymphodepletion therapy.
23. Allogenic stem cell transplantation within last two months or GvHD requiering systemic immunosuppressive therapy.
24. Vaccination with live viruses within 2 weeks prior to lymphodepletion therapy.
25. Major surgery within 28 days (prior to start of TM123 infusion)
26. Other malignancy requiring active therapy, but adjuvant endocrine therapy is allowed.
27. Treatment with any investigational drug substance or experimental therapy within 4 weeks or 5 half-lives (whatever is shorter) of the substance prior to the day of apheresis
28. Prior treatment with gene therapy products unless approved by the sponsor.
29. Use of checkpoint inhibitors within 5 half-lives of the respective substance.
30. Pregnatn or breastfeeding women.
31. Currently significant psychologic disorder, including substance abuse.
32. Known history of human immunodeficiency virus (HIV) or human T-lymphotropic virus (HTLV) or active/chronic infection with hepatitis C virus (HCV) or hepatitis B virus (HBV).
33. Any significant autoimmune disease requiring systemic immunosuppressive therapy or that may otherwise, in the Investigator''s opinion, interfere with participation in the trial, or documented presence of autoantibodies against La/SS-B.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2020-01-28 (Actual); Primary Completion 2025-04-11 (Actual); Study Completion 2025-04-11 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability | Infusion period of TM123 (up to 20 days) + 7 days resp. 14 days in patients with complete blast clearance during the IC or until Safety Follow-up 1 (infusion period of TM123 + 28 days + 3 months)
  Incidence and intensity of adverse events graded according to CTCAE V5.0 with the exception of CRS and ICANS graded according to Lee et al. 2014 and Lee et al. 2019 respectively
Recommended phase 2 dose (RP2D) | Infusion period of TM123 (up to 20 days) + 7 days or + 14 days in patients with complete blast clearance)
  Establishing recommended phase 2 dose (RP2D) and schedule
Response | Infusion period of TM123 (up to 20 days) + 7 days or + 14 days in patients with complete blast clearance)
  Complete remission (CR, CRh, CRi, CRMRDneg, CRMRDpos) and partial remission (PR) at any time point and duration of responses

SECONDARY OUTCOMES:
Establishing recommended phase 2 dose (RP2D) | DLT period (infusion period of TM123 (up to 20 days) + 7 days or + 14 days in patients with complete blast clearance)
  The RP2D will be determined based on MTD, all available efficacy data, and all available safety data, including information derived from additional treatment cycles.
Complete (CR, CRh, CRi ) and partial remission (PR) | until fifteen years after last UniCAR02-T administration
  CR: Bone marrow blasts < 5%, absence of extramedullary disease, absolute neutrophil count > 1 Gpt/L and platelet count > 100 Gpt/L. Level of MRD should be measured in patients achieving CR in case as suitable marker exists.
  CRi: All criteria for CR except residual thrombocytopenia (platelets < 100 Gpt/L) and/or neutropenia (absolute neutrophil count < 1 Gpt/L).
  PR: All hematological criteria for CR with bone marrow blasts 5-25% and decrease of pre-treatment bone marrow blast percentage by at least 50 %.
Disease stabilization (DS) | until fifteen years after last UniCAR02-T administration
  Reduction of blast percentage by 25% compared to baseline without normalization of peripheral blood counts to levels not qualifying for PR or CR.
Best response rate | until fifteen years after last UniCAR02-T administration
  The best observed response during observational period. Response states are ordered descending as follows: CR > CRi > PR > DS > refractory disease.
Progression free survival (PFS) | until fifteen years after last UniCAR02-T administration
  The time from first treatment with TM123 and UniCAR02-T until disease progression or death. If no progress of death was observed during the observational period, the patient's progression free survival time will be censored on the date the patient was last seen progression-free and alive.
Overall survival (OS) | until fifteen years after last UniCAR02-T administration
  The number of days between the first study drug administration and death from any cause. If death was not observed during the observational period, the patient's overall survival time will be censored on the date the patient was last seen alive.
Toxicity and efficacy in repeated cycles of TM123 administration | duration of consolidation cycle treatment
  Patients who tolerate TM123 and UniCAR02-T without DLT and achieve a clinical benefit are candidates for consolidation cycles

CONTACTS AND LOCATIONS:
Locations (10):
- Germany (8):
  - Universitätsklinikum Ulm, Ulm, Baden-Wurttemberg
  - Klinikum der Universität München, Munich, Bavaria
  - Universitätsklinikum Würzburg, Würzburg, Bavaria
  - Philipps-Universität Marburg, Marburg, Hesse
  - Uniklinik RWTH Aachen, Aachen, North Rhine-Westphalia
  - Universitätsklinikum Dresden, Dresden, Saxony
  - Universitätsklinikum Leipzig, Leipzig, Saxony
  - Universitätsklinikum Hamburg-Eppendorf, Hamburg
- Netherlands (2):
  - Erasmus University Medical Center, Rotterdam, Gelderland
  - Universitair Medisch Centrum Groningen, Groningen, GZ

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Loff S, Dietrich J, Meyer JE, Riewaldt J, Spehr J, von Bonin M, Grunder C, Swayampakula M, Franke K, Feldmann A, Bachmann M, Ehninger G, Ehninger A, Cartellieri M. Rapidly Switchable Universal CAR-T Cells for Treatment of CD123-Positive Leukemia. Mol Ther Oncolytics. 2020 Apr 29;17:408-420. doi: 10.1016/j.omto.2020.04.009. eCollection 2020 Jun 26. PMID 32462078